CLINICAL TRIAL: NCT02600910
Title: Natural History of Shoulder Pathology in Manual Wheelchair Users
Acronym: NHSSI
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Mayo Clinic (Other); West Virginia University (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0127; 15-004974 (Other: Mayo Clinic)
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Paraplegia; Spinal Cord Injuries; Shoulder Pain; Tendinopathy
Keywords: Manual Wheelchair; Shoulder injury; Shoulder function; rotator cuff; Tendinopathy; Spinal cord injury; Shoulder pain; Shoulder impingement
MeSH Terms: conditions — Paraplegia; Spinal Cord Injuries; Shoulder Pain; Tendinopathy; Shoulder Injuries; Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Manual Wheelchair User Cohort: Physical Exam. Screening exam performed by a licensed physical therapist to confirm inclusion/exclusion criteria.
  Assessment of Shoulder Function in Everyday Life. Shoulder motion & hand loading data will be collected over a few days, twice per yr for 3-5 yrs in home & community environment.
  Magnetic Resonance Imaging (MRI) of Shoulders. Imaging will use standard clinical protocol once per yr for 3-5 yrs.
  Shoulder Strength Testing. Once per yr for 3-5 yrs. Additional Variables. Updated demographic info will be collected yearly including but not limited to weight, chair type, health status, and job type.
- Matched Able-bodied Cohort: Physical Exam. Screening exam performed by a licensed physical therapist to confirm inclusion/exclusion criteria.
  Assessment of Shoulder Function in Everyday Life. Shoulder motion & hand loading data will be collected over a few days, twice per yr for 3-5 yrs in home & community environment.
  Magnetic Resonance Imaging (MRI) of Shoulders. Imaging will use standard clinical protocol once per yr for 3-5 yrs.
  Shoulder Strength Testing. Once per yr for 3-5 yrs. Additional Variables. Updated demographic info will be collected yearly including but not limited to weight, health status, and job type.

SUMMARY:
Over 300,000 people in the United States have spinal cord injuries and many use manual wheelchairs for mobility. Most manual wheelchair users will develop shoulder injuries and pain that greatly affect quality of life and level of independence. Understanding when shoulder disease starts in manual wheelchair users and which daily activities contribute to the disease will provide necessary evidence for effective primary prevention methods to inhibit the development of further disability. Our central hypothesis is that the development of shoulder disease in manual wheelchair users will be strongly associated with the cumulative exposure to elevated shoulder postures combined with high upper body loading.

DETAILED DESCRIPTION:
Of the 1.7 million wheelchair users in the United States (US), 90 percent, or 1.5 million persons use manual wheelchairs (MWCs). People with traumatic and non-traumatic spinal cord injuries (SCI) make up approximately 20% of the MWC users, and 12,000 new traumatic SCIs occur every year. While MWCs are immediately available and enable independence, 63% of MWC users will have one or multiple rotator cuff tears after decades of MWC use as compared to 15% of age-matched able-bodied adults. A crucial gap in knowledge exists in understanding how the shoulder of MWC users functions from an almost permanent seated position as an agent for mobility, weight bearing, and hand grasping; and how this altered function translates to longitudinal shoulder health decline.

The objective of this application is to define the longitudinal components of the early phase (before chronic symptom onset) of shoulder health decline specific to new MWC users by characterizing the exposure to altered shoulder function and the associated MRI signs of early onset of shoulder pathology. The investigators propose to: (Aim 1) quantify shoulder joint motion and loading in the real world over 3 years in 50 new MWC users and a matched able-bodied cohort; (Aim 2) define early, preclinical changes on shoulder MRI specific to the MWC users, over 3 years, in comparison to the matched cohort; and (Aim 3) identify specific exposure measures as risk factors for early changes on MRI in the MWC users. Three central and novel aspects of this proposal will pave the way for targeting primary prevention: (1) characterizing the altered shoulder function in new MWC users in the real world with hardware and instrumentation suitable for multiple, day long collections, (2) defining the early, preclinical pattern of disease in users compared to a matched able-bodied cohort, and (3)investigating the combined effect of shoulder motion and loading and its relationship to the incidence of shoulder pathology.

Successful completion of this project will define how the shoulder responds to MWC use (Aim 1), identify the MWC-specific pattern of shoulder disease on MRI (Aim 2), and determine how altered shoulder function has contributed to shoulder health decline (Aim 3). This work provides the foundation for understanding the relative impact of shoulder elevation and loading in shoulder health decline. Additionally, this work provides the first building block in defining the complete natural history of shoulder disease in MWC users. The investigators expect the overall impact to be a powerful influence on environmental and assistive technology redesign, post-SCI rehabilitation practices, insurance reimbursement for shoulder health-preserving equipment, and understanding shoulder pathology in the general population.

ELIGIBILITY:
Inclusion Criteria:

Group1 (Manual Wheelchair User Cohort):

* Participants with traumatic or non-traumatic spinal cord injury who have begun using a MWC within 12 months of enrollment
* 18 - 70 years of age
* Use of a manual wheelchair as the primary mode of mobility
* Functional upper extremity range of motion
* Willingness to participate in study
* Ability to return to receive shoulder MRI 1-3 times/year , and once per year receive physical exam, and strength assessments.

Group 2 (Matched Able-bodied Cohort):

* 18-70 years of age
* Able to walk independently with no reliance on an orthotic, prosthetic, or gait aid
* Functional upper extremity range of motion
* Willingness to participate in study
* Ability to receive shoulder MRI 1-3 times/year, and once per year receive physical exam, and strength assessments.

Exclusion Criteria:

Group1 (Manual Wheelchair User Cohort):

• Previous diagnosis of bilateral shoulder tendon tears prior to spinal cord injury or suspected tendon tears with physical exam

Group 2 (Matched Able-bodied Cohort):

* Any documented musculoskeletal or neurological disorders that would be expected to impact shoulder health or change ability to walk independently
* Previous diagnosis of shoulder tears prior to enrollment or suspected tendon tears with physical exam

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 new manual wheelchair users with traumatic or non-traumatic spinal cord injuries (SCI) will be recruited & consented during the first 2 years of this project. Subjects will be recruited at sites that treat & rehabilitate people with acute SCI. SE MN & neighboring states will be the 1st regions of recruitment. The inclusion and exclusion criteria were chosen to include a sample of the population of people with new SCIs who will use MWCs as their primary mode of mobility inside and outside the home. For 25 SCI participants, an age, sex, and activity level able-bodied matched participant will be recruited from the SE MN area.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Participant completion of MRI and Field measurements after 3 to 5 years follow-up. | 3-5 years
  Investigators will use the standardized MRI Assessment of the shoulder guide to assess shoulder pathology and compare baseline shoulder condition on MRI to yearly follow-up. For the purposes of grading, pathology aside from rotator cuff tears will be assessed on an ordinal scale from 0-3 with 0 indicating no abnormality, 1 mild, 2 moderate, and 3 severe. Field measurements will be used to determine changes in upper extremity motion and loading from baseline across 3-5 years of follow-up.

SECONDARY OUTCOMES:
Development of the Conceptual Model of Preclinical Natural History of Shoulder Health Decline. | 3-5 years
  Investigators will model the preclinical phase of shoulder health decline based on the Natural History of Disease. The exposure variables are defined by the upper extremity motion and loading, and the biological onset of the disease and pattern of disease development will be defined with the MRI findings of pathology type, location, and severity. Using regression techniques, an exposure-response relationship will be defined.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Morrow, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
This will be decided further into the study.